CLINICAL TRIAL: NCT00976131
Title: Phase I Randomized, Placebo-Controlled, Cross-Over, Dose-Finding Pharmacokinetic Study of CoQ10 During One Cycle of Doxorubicin Treatment for Breast Cancer
Brief Title: Study of CoQ10 During One Cycle of Doxorubicin Treatment for Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AAAD8521
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Early Stage Breast Cancer; Complementary and Alternative Medicine; CAM
MeSH Terms: conditions — Breast Neoplasms | interventions — coenzyme Q10; Doxorubicin; liposomal doxorubicin; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A Placebo (Placebo Comparator): Patients will begin taking their study pills (CoQ10) on the morning of Cycle 2 Day 3 (11-15 days prior to Cycle 3), and will continue taking the study pills through the morning of their Cycle 3 infusion (Day 1 Cycle 3). Patients will then be crossed-over to the alternative condition. On the morning of Cycle 3 Day 3, patients will begin taking their study pills (CoQ10 placebo) and will continue taking the study pills through the morning of their Cycle 4 infusion (Day 1 Cycle 4).
  Infusion will be standard of care chemotherapy with doxorubicin and cyclophosphamide.
  Interventions: Drug: CoQ10; Other: CoQ10 Placebo; Drug: Doxorubicin; Drug: Cyclophosphamide
- Arm B CoQ10 (Experimental): Patients will begin taking their study pills (CoQ10 placebo) on the morning of Cycle 2 Day 3 (11-15 days prior to Cycle 3), and will continue taking the study pills through the morning of their Cycle 3 infusion (Day 1 Cycle 3). Patients will then be crossed-over to the alternative condition. On the morning of Cycle 3 Day 3, patients will begin taking their study pills (CoQ10) and will continue taking the study pills through the morning of their Cycle 4 infusion (Day 1 Cycle 4).
  Infusion will be standard of care chemotherapy with doxorubicin and cyclophosphamide.
  Interventions: Drug: CoQ10; Other: CoQ10 Placebo; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: CoQ10 — Capsules taken daily for two weeks prior to Cycle 3 chemotherapy infusion OR Capsules taken daily for two weeks prior to Cycle 4 infusion.
  Dose Level 1: 300mg/d CoQ10 (2 capsules) Dose Level 2: 600mg/d CoQ10 (4 capsules) Dose Level 3: 1200mg/d CoQ10 (8 capsules)
  Other Names: Coenzyme Q10
Other: CoQ10 Placebo — Capsules taken daily for two weeks prior to Cycle 3 chemotherapy infusion OR Capsules taken daily for two weeks prior to Cycle 4 infusion.
  Dose Level 1: 300mg/d placebo (2 capsules) Dose Level 2: 600mg/d placebo (4 capsules) Dose Level 3: 1200mg/d placebo (8 capsules)
  Other Names: Coenzyme Q10 Placebo
Drug: Doxorubicin — Standard of care chemotherapy medication used to treat cancer.
  Other Names: Doxil
Drug: Cyclophosphamide — Standard of care chemotherapy medication used to treat cancer.
  Other Names: Cytoxan

SUMMARY:
This research study hopes to examine the effects of Coenzyme Q10 on doxorubicin (Adriamycin) metabolism during breast cancer treatment.

DETAILED DESCRIPTION:
Doxorubicin is a lifesaving breast cancer treatment. However, approximately 3-20% of women who receive doxorubicin treatment experience some damage to their heart muscle. Coenzyme Q10 is a fat soluble antioxidant dietary supplement that may protect against this heart damage during doxorubicin treatment. It is unknown how Coenzyme Q10 may interact with doxorubicin. This study will assess the effects of Coenzyme Q10 on doxorubicin metabolism.

This is a phase I randomized, placebo-controlled, cross-over pharmacokinetic and dose-finding study to assess the safety of CoQ10 during doxorubicin treatment for breast cancer. Safety will be assessed by measuring 1) intra-patient differences in doxorubicin and its active metabolites, with and without CoQ10, and 2) adverse events. The investigator hypothesizes that CoQ10 administration during doxorubicin treatment is safe and will not affect doxorubicin active metabolites. Using three dose levels of CoQ10, the maximum tolerated dose (MTD) will be determined by assessing change in doxorubicin concentration (area under the curve (AUC), change in peak concentration levels (Cmax)), and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of early stage breast cancer (stage I, II, or III);
* Scheduled to receive at least four rounds of dose dense doxorubicin therapy in the neoadjuvant or adjuvant setting;
* No other history of prior chemotherapy, radiation, or hormonal therapy in the previous 5 years;
* For women receiving adjuvant therapy, single lumen implanted venous access device (i.e. single port) for unilateral cancer and double lumen implanted venous access device (i.e. double port) for bilateral breast cancer
* Age 21 years or older;
* ECOG performance status ≤ 2 (Karnofsky > 60%);
* Normal organ and marrow function defined as: Leukocytes ≥ 3,000/uL, Absolute neutrophils count (ANC) ≥ 1,500/uL at baseline, Platelets ≥ 100,000/uL, Total bilirubin ≤ 1.5 X normal institutional limits, AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional ULN, Serum creatinine within normal institutional limits;
* Left ventricular ejection fraction > 55%;
* No history of CoQ10 supplement use within 30 days of initiating study drug;
* No uncontrolled or significant co-morbid illness;
* Not pregnant, not breastfeeding, and not planning on becoming pregnant during the course of the study;
* Willingness to comply with all study intervention and follow-up procedures;
* Ability to speak English or Spanish; and
* Ability to provide informed consent.

Exclusion Criteria:

* Inability to understand or an unwillingness to sign a written informed consent document;
* Any significant toxic side effects related to first or second dose of doxorubicin/cyclophosphamide chemotherapy or biologic therapy that did not resolve to less than a CTCAE 3.0 grade 3 non-hematological toxicity;
* Currently using any investigational agent;
* Unstable or severe intercurrent medical condition that, in the opinion of the investigator, might interfere with the participant's ability to follow the protocol or achieve study objectives;
* Psychological or sociological conditions, addictive disorders, or family problems that would preclude adherence with study drug or compliance with the protocol
* Women who report pregnancy, are breast feeding, or have a positive pregnancy test;
* Use of CoQ10 supplement use within 30 days of initiating study drug;
* Use of over-the-counter nutritional vitamin greater than 5x RDA;
* Fish allergy (due to fish-based softgel shell);
* Currently taking FDA cardioprotective drugs, such as Zinecard (dexrazoxane);
* History of chronic hepatitis B, hepatitis C, and HIV infection;
* Problems swallowing oral medications due to prolonged emesis, mucositis, esophageal dysfunction, etc.; and,
* Currently taking any form of antioxidant supplements while on study.
* Use of warfarin.
* Kosher (due to fish-based softgel shell)
* Dietary restriction of tilapia (due to tilapia fish-based softgel shell)
* Titanium Dioxide allergy (due to the opaque coloring used in the softgel).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2012-09-30 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of CoQ10 that does not alter the pharmacokinetics of doxorubicin | At the end of Cycle 4 Day 2 (each cycle is 21 days)
  To test increasing doses on different groups of people until the highest dose with acceptable side effects is found.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Greenlee, ND, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Greenlee H, Crew KD, Maurer M, Kalinsky K, Cremers S, Naini A, Tsai WY, Shi Z, Brogan F, Hershman DL. Phase I Randomized, Placebo-Controlled, Cross-Over Dose-Finding Study of Coenzyme Q10 on Doxorubicin Pharmacokinetics during Breast Cancer Treatment. Integr Cancer Ther. 2025 Jan-Dec;24:15347354251388014. doi: 10.1177/15347354251388014. Epub 2025 Nov 19. PMID 41261512